CLINICAL TRIAL: NCT01294592
Title: Comparative Efficacy of DuodartTM Versus Watchful Waiting With Step-up Therapy to Tamsulosin in the Management of Treatment naïve Men With Symptomatic BPH
Brief Title: Comparative Efficacy of Dutasteride Plus Tamulosin With Lifestyle Advice Versus Watchful Waiting Plus Lifestyle Advice in the Management of Treatment naïve Men With Moderately Symptomatic Benign Prostatic Hyperplasia and Prostate Enlargement
Acronym: CONDUCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114615
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tamsulosin

ARMS (2):
- Dutasteride plus tamsulosin (Active Comparator): Dutasteride plus tamsulosin arm + lifestyle advice
  Interventions: Drug: Dutasteride plus tamsulosin
- Watchful waiting with escalation to tamsulosin (Experimental): Watchful waiting with escalation to tamsulosin
  Interventions: Drug: tamsulosin

INTERVENTIONS:
Drug: Dutasteride plus tamsulosin — Take 1 capsule daily
  Arms: Dutasteride plus tamsulosin
Drug: tamsulosin — Take 1 capsule daily when escalation criteria met
  Arms: Watchful waiting with escalation to tamsulosin

SUMMARY:
Study FDC114615 is a two year, multi-centre, randomised, open-label trial to assess the efficacy of Dutasteride plus tamsulosin when compared to the standard practice of watchful waiting, with a defined escalation to tamsulosin in treatment naive men with symptomatic benign prostate hyperplasia (BPH).

Once consented, each subject will undergo screening procedures to ensure the prostate volume and post void residual are within eligible range. If all entry criteria are met, subjects will be randomised (1:1) to receive Dutasteride plus tamsulosin with lifestyle advice or watchful waiting, with lifestyle advice, with a defined escalation to tamsulosin. Escalation will be initiated when no improvement from baseline is scored using the International Prostate Symptom Score (version 2) (IPSS) questionnaire.

After randomisation, the subjects return to site at one month, then every 13 weeks until two years of treatment is complete or they are withdrawn. Key assessments, such as Adverse Events (AE's) and concomitant medication monitoring and completion of the quality of life questionnaires are performed at each visit and the data recorded.

DETAILED DESCRIPTION:
This will be a European, multicentre, randomised, open-label, parallel group study. The aim of the study is to investigate whether Dutasteride plus Tamulson treatment with lifestyle advice is more effective than watchful waiting treatment plus lifestyle advice plus step-up therapy with tamsulosin for improvement of symptoms and Acte Urinary Retention (AUR) and BPH-related prostatic surgery, in older men (≥50 yrs), with moderate symptoms of BPH (IPSS 8-19), enlarged prostates (≥30cc) and Prostate Specific Antigen (PSA) ≥1.5ng/mL.

Data from all participating centres will be pooled prior to analysis. Investigative centres will be pooled a priori into clusters based on geographic location; these clusters may be used in analyses to adjust for site effects. Clusters will be defined once all investigative centres have been identified and randomisation has been completed.

Subjects will be screened for inclusion into the study and eligible subjects will be randomised by investigative centre. Subjects will be allocated to one of two treatment groups, according to a pre-determined randomisation schedule (in a 1:1 ratio):

* Dutasteride plus tamsulosin once daily plus lifestyle advice.
* Watchful waiting plus lifestyle advice. Escalation to tamsulosin 0.4 mg once daily at any visit from Week 4 if any IPSS measurement shows no improvement or worsening from baseline. At any study visit, if the IPSS is the same or greater than the baseline value for that subject, tamsulosin 0.4 mg once daily will be initiated. If tamsulosin is initiated, it will be continued for the remainder of the study unless the subject elects to withdraw from the study. Initiation of tamsulosin will be recorded in the electronic case report form (eCRF.) Subjects will self-administer study medication once daily for up to 104 weeks, (up to 100 weeks for those on tamsulosin). Subjects will return to the clinic at 4 weeks post-randomisation and then at 13-week intervals post-randomisation during the 2-year treatment period (i.e. at 4, 13, 26, 39, 52, 65, 78, 91 and 104 weeks) for the assessments listed as in Appendix 1 Time and Events Schedule.

Approximately 760, treatment naive men with symptomatic BPH will be randomised into the study in order to achieve at least 592 evaluable subjects. 380 into the Dutasteride plus tamsulosin with lifestyle advice arm and 380 into the watchful waiting plus lifestyle advice arm.

Treatment naïve is defined as a man that has recently been diagnoses with BPH whom has received no prescribed therapeutic treatment. For example, medicines such as 5 α-reductase inhibitors (5-ARIs) or invasive procedures such as transurethral resection of the prostate (TURP) prescribed to directly treat the BPH symptoms are considered therapeutic treatments. As per the entry criteria, phytotherapy is allowed unless it was performed less than two weeks prior to the screening visit.

The anticipated recruitment period will be approximately 6 months. The study will be conducted in approximately 8 countries within Europe.

ELIGIBILITY:
* Males aged ≥50 years.
* A confirmed clinical diagnosis of BPH.
* International Prostate Symptom Score (IPSS) 8-19 at Visit 1 (screening).
* Prostate volume ≥30 cc (by transrectal ultrasonography; TRUS).
* Total serum prostate specific antigen (PSA) ≥1.5 ng/mL at Visit 1 (screening).
* Willing and able to give signed written informed consent and comply with study procedures.
* Fluent and literate in local language with the ability to read, comprehend and record information on the IPSS and BII questionnaires.
* Able to swallow and retain oral medication.
* Willing and able to participate in the study for the full 2 years.
* Men with a female partner of childbearing potential must either agree to use effective contraception or have had a prior vasectomy. Contraception must be used from 2 weeks prior to administration of the first dose of study treatment until at least 5 half-lives for the drug plus 3 months to allow clearance of any altered sperm after the last dose of study treatment.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Note: If total serum PSA is >4 ng/mL and unless PSA value has been stable for at least the past 2 years, the investigator should make every appropriate effort to exclude the possibility of prostate cancer, e.g. further Digital rectal examination (DRE), review TRUS taken within previous month, consider 8-12 core prostate biopsy in accordance with routine clinical practice

Exclusion Criteria:

* Subjects meeting any of the following criteria must not be enrolled in the study:
* Total serum PSA >10.0 ng/mL at Visit 1 (screening).
* History or evidence of prostate cancer (e.g. positive biopsy or ultrasound within the previous 6 months, suspicious DRE and/or rising PSA).

Excluded medication and therapies Current or any prior use of the following prohibited medications

* a 5α-reductase inhibitor (finasteride or dutasteride),
* anti-cholinergics (e.g. oxybutynin, propantheline)
* an alpha-adrenoreceptor blocker (i.e. indoramin, prazosin, terazosin, tamsulosin, alfuzosin and doxazosin) for BPH or Lower urinary tract symptoms (LUTS)
* any drugs with anti-androgenic properties (e.g. spironolactone, flutamide, bicalutamide, cimetidine, ketoconazole, progestational agents) within the previous 6 months.
* any drugs noted for gynaecomastia effects, or could affect prostate volume, within 6 months of the Visit 1
* any investigational or marketed study drug within 30 days or 5 half-lives, (whichever is longer), preceding the first dose of study treatment.

Current use of:

* any alpha-adrenoreceptor blocker (i.e. indoramin, prazosin, terazosin, tamsulosin, alfuzosin and doxazosin)
* anabolic steroids.
* drugs known or thought to have an interaction with tamsulosin, e.g. cimetidine and warfarin.
* Use of phytotherapy for BPH within 2 weeks prior to Visit 1 (screening) and/or predicted to need phytotherapy during the study.

Have a known (immediate or delayed) hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study medication or excipients that, in the opinion of the Investigator or GlaxoSmithKline contraindicates their participation.

Recent Medical Procedures

* Previous prostatic surgery (including TURP, balloon dilatation, thermotherapy and stent replacement) or other invasive or minimally invasive procedures to treat BPH.
* History of flexible/rigid cystoscopy or other instrumentation of the urethra within 7 days prior to Visit 1 (screening). Catheterisation (<10F) is acceptable with no time restriction.

Medical history

* History of AUR within 3 months prior to Visit 1 (screening).
* Post-void residual volume >250 mL (suprapubic ultrasound) at Visit 1 (screening)..
* Any causes other than BPH, which may in the judgement of the investigator, result in urinary symptoms or changes in flow rate (e.g. neurogenic bladder, bladder neck contracture, urethral stricture, bladder malignancy, acute or chronic prostatitis, or acute or chronic urinary tract infections).
* History of 'first dose' hypotensive episode on initiation of alpha-1-adrenoreceptor antagonist therapy for hypertension.
* History of postural hypotension, dizziness, vertigo or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
* History of breast cancer or clinical breast examination finding of unclear origin or suggestive of malignancy.
* History of hepatic impairment or abnormal liver function tests at Visit 1 (screening). (defined as Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) or alkaline phosphatase >2 times the Upper limit of normal (ULN) , or total bilirubin >1.5 times the ULN, (unless associated with predominantly indirect bilirubin elevation or Gilbert's syndrome).
* History of renal insufficiency, or serum creatinine >1.5 times the upper limit of normal at Visit 1 (screening)..
* Prior history of malignancies (other than basal cell carcinoma or squamous cell carcinoma of the skin) within the past 5 years. Subjects who have had no evidence of the malignancy for ≥5 years are eligible.
* History of any illness (including psychiatric) that in the opinion of the investigator might confound the results of the study or poses additional risk to the subject.
* Any unstable, serious co-existing medical condition(s) including, but not limited to, myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to Screening visit; uncontrolled diabetes or peptic ulcer disease which is uncontrolled by medical management.
* History or current evidence of drug or alcohol abuse within the previous 12 months.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator or GSK Medical Monitor.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2010-12-22 (Actual); Primary Completion 2013-10-17 (Actual); Study Completion 2013-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (75):
- France (14):
  - GSK Investigational Site, Aigrefeuille-sur-Maine
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Corsept
  - GSK Investigational Site, La Montagne
  - GSK Investigational Site, La Rochelle
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Le Temple-de-Bretagne
  - GSK Investigational Site, Mûrs-Erigné
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nieul-sur-Mer
  - GSK Investigational Site, Sautron
  - GSK Investigational Site, Thouars
  - GSK Investigational Site, Tiercé
  - GSK Investigational Site, Vihiers
- Germany (13):
  - GSK Investigational Site, Aichach, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Hagenow, Brandenburg
  - GSK Investigational Site, Oranienburg, Brandenburg
  - GSK Investigational Site, Strausberg, Brandenburg
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Buchholz, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Hettstedt, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Eisleben Lutherstadt
- Greece (6):
  - GSK Investigational Site, Argos
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Rhodes
  - GSK Investigational Site, Thessaloniki
- Italy (10):
  - GSK Investigational Site, Vasto (CH), Abruzzo
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Avellino, Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, San Fermo Della Battaglia (CO), Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Pisa, Tuscany
- Netherlands (7):
  - GSK Investigational Site, Doetinchem
  - GSK Investigational Site, Maarssen
  - GSK Investigational Site, Sneek
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Voerendaal
  - GSK Investigational Site, Wildervank
  - GSK Investigational Site, Winterswijk
- Romania (2):
  - GSK Investigational Site, Arad
  - GSK Investigational Site, Bucharest
- Spain (15):
  - GSK Investigational Site, Alava
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Coslada
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Fuenlabrada (Madrid)
  - GSK Investigational Site, Galdakano
  - GSK Investigational Site, Getafe
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Mendaro, Guipuzcoa
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
- United Kingdom (8):
  - GSK Investigational Site, Chalfont St Giles, Buckinghamshire
  - GSK Investigational Site, Sandbach, Cheshire
  - GSK Investigational Site, Bath
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Broadway, Fleetwood
  - GSK Investigational Site, Chadderton, Oldham
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, High Heaton, Newcastle Upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment-naïve men with symptomatic benign prostatic hyperplasia (BPH) meeting eligibility criteria were enrolled and were randomized in a 1:1 ratio to receive dutasteride plus tamsulosin once daily plus lifestyle advice or watchful waiting plus lifestyle advice.
Groups:
- Dutasteride Plus Tamsulosin: Participants received a combination of dutasteride 0.5 milligrams (mg) plus tamsulosin 0.4 mg plus lifestyle advice for 24 months.
- Watchful Waiting All: Escalated Yes and No: All participants were given lifestyle advice. If any International Prostate Symptom Score (IPSS) was the same or greater than the Baseline value at any study visit (post-randomization), participants received tamsulosin 0.4 mg once daily (Watchful Waiting Escalated=Yes). Tamsulosin was continued until the end of the study unless the participant elected to withdraw from the study. If participants did not receive tamsulosin, they were not classified as escalated (Watchful Waiting Escalated=No).
Period: Overall Study
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No
Started | 369 | 373
Completed | 292 | 300
Not Completed | 77 | 73
Not completed — Adverse Event | 28 | 13
Not completed — Lack of Efficacy | 7 | 5
Not completed — Protocol Violation | 1 | 7
Not completed — Lost to Follow-up | 7 | 9
Not completed — Physician Decision | 6 | 11
Not completed — Withdrawal by Subject | 28 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No | Total
Number analyzed (Participants) | 369 | 373 | 742
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.3 (7.78) | 66.2 (7.34) | 66.2 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 369 | 373 | 742
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 357 | 363 | 720
  White - Arabic/North African Heritage | 4 | 2 | 6
  African American/African Heritage | 0 | 2 | 2
  Mixed Race | 0 | 1 | 1
  Missing | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total International Prostate Symptom Score (IPSS) at Months 1, 3, 6, 9, 12, 15, 18, 21, and 24 Using the Last Observation Carried Forward (LOCF) Approach
Description: The IPSS questionnaire is a 7-item self-administered questionnaire designed to quantify the following urinary symptoms: Question 1 (Q1), incomplete emptying; Q2, frequency; Q3, intermittency; Q4, urgency; Q5, weak stream; Q6, straining; Q7, nocturia. It has an additional, independent eighth question to assess change in BPH-related health status (BHS) and quality of life. BHS scores range from 0 to 6, where 0 indicates "delighted" and 6 indicates "terrible." The 7 items in the IPSS questionnaire quantitatively measure the level of urinary symptoms reported as a total IPSS. The total IPSS (sum of the first 7 items) can range from 0 to 35: mild (0 to 7), moderate (8 to 19), or severe (20 to 35). Change from Baseline in IPSS total score was calculated as the Month 24 value minus the Baseline value. LOCF analysis involves bringing forward the last non-missing post-Baseline assessment for a participant with missing data and/or for a participant who discontinued from the study.
Time Frame: Baseline and Months 1, 3, 6, 9, 12, 15, 18, 21, and 24
Population: Intent-to-Treat (ITT) Population: all randomized participants regardless of whether or not treatment was administered. Any participant who received a treatment randomization number was considered to have been randomized. Participants with data available at the specified time point or using LOCF (post-Baseline) were summarized.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No
Number analyzed (Participants) | 359 | 368
Scores on a scale
  Month 1, n=358, 367 | -3.2 (0.21) | -0.9 (0.20)
  Month 3, n=359, 368 | -4.5 (0.22) | -2.4 (0.22)
  Month 6, n=359, 368 | -4.6 (0.23) | -3.2 (0.22)
  Month 9, n=359, 368 | -5.1 (0.22) | -3.6 (0.22)
  Month 12, n=359, 368 | -5.2 (0.23) | -3.6 (0.23)
  Month 15, n=359, 368 | -5.2 (0.25) | -3.6 (0.24)
  Month 18, n=359, 368 | -5.1 (0.25) | -3.3 (0.25)
  Month 21, n=359, 368 | -5.5 (0.25) | -3.6 (0.24)
  Month 24, n=359, 368 | -5.4 (0.25) | -3.6 (0.25)
Statistical Analysis 1: Comparison: Dutasteride Plus Tamsulosin vs Watchful Waiting All: Escalated Yes and No; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Month 1; Values are based on t-tests from the general linear model; Adjusted Mean Difference = -2.2, 95% CI 2-sided [-2.8 to -1.7], Standard Error of Mean 0.28 — Estimates are based on the adjusted means from the general linear model: Change from Baseline = Treatment + Cluster + Baseline Value. The adjusted mean difference is based on dutasteride plus tamsulosin minus Watchful Waiting All
Statistical Analysis 2: Comparison: Dutasteride Plus Tamsulosin vs Watchful Waiting All: Escalated Yes and No; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Month 3; Values are based on t-tests from the general linear model; Adjusted Mean Difference = -2.1, 95% CI 2-sided [-2.7 to -1.5], Standard Error of Mean 0.31 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dutasteride Plus Tamsulosin vs Watchful Waiting All: Escalated Yes and No; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Month 6; Values are based on t-tests from the general linear model; Adjusted Mean Difference = -1.5, 95% CI 2-sided [-2.1 to -0.9], Standard Error of Mean 0.31 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Dutasteride Plus Tamsulosin vs Watchful Waiting All: Escalated Yes and No; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Month 9; Values are based on t-tests from the general linear model; Adjusted Mean Difference = -1.6, 95% CI 2-sided [-2.2 to -1.0], Standard Error of Mean 0.31 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Dutasteride Plus Tamsulosin vs Watchful Waiting All: Escalated Yes and No; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Month 12; Values are based on t-tests from the general linear model; Adjusted Mean Difference = -1.6, 95% CI 2-sided [-2.2 to -1.0], Standard Error of Mean 0.32 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Dutasteride Plus Tamsulosin vs Watchful Waiting All: Escalated Yes and No; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Month 15; Values are based on t-tests from the general linear model; Adjusted Mean Difference = -1.6, 95% CI 2-sided [-2.3 to -1.0], Standard Error of Mean 0.34 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Dutasteride Plus Tamsulosin vs Watchful Waiting All: Escalated Yes and No; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Month 18; Values are based on t-tests from the general linear model; Adjusted Mean Difference = -1.7, 95% CI 2-sided [-2.4 to -1.0], Standard Error of Mean 0.35 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Dutasteride Plus Tamsulosin vs Watchful Waiting All: Escalated Yes and No; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Month 21; Values are based on t-tests from the general linear model; Adjusted Mean Difference = -1.9, 95% CI 2-sided [-2.5 to -1.2], Standard Error of Mean 0.34 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Dutasteride Plus Tamsulosin vs Watchful Waiting All: Escalated Yes and No; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Month 24; Values are based on t-tests from the general linear model; Adjusted Mean Difference = -1.8, 95% CI 2-sided [-2.5 to -1.2], Standard Error of Mean 0.34 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With Change From Baseline in the Indicated Improvement Categories in the IPSS at Months 1, 3, 6, 9, 12, 15, 18, 21, and 24 Using the LOCF Approach
Description: Symptom improvement was assessed using IPSS categorical changes from Baseline. Change from Baseline categories were summarized by treatment group using five improvement levels: >=1 point through >=5 points. IPSS percent change from Baseline was summarized using seven improvement levels: >0 percent, >=10 percent, >=20 percent, >=25 percent, >=30 percent, >=40 percent, and >=50 percent. Change in IPSS from Baseline was analysed using the LOCF method and is summarized for the following categories: >=2 points, >=3 points, and percent change >=25. The 7 items in the IPSS questionnaire quantitatively measure the level of urinary symptoms reported as a total IPSS. The total IPSS (sum of the first 7 items) can range from 0 to 35: mild (0 to 7), moderate (8 to 19), or severe (20 to 35).
Time Frame: Baseline and Months 1, 3, 6, 9, 12, 15, 18, 21, and 24
Population: ITT Population. Participants with data available at the specified time point or using LOCF (post-Baseline) were summarized. LOCF analysis involves bringing forward the last non-missing post-Baseline assessment for a participant with missing data and/or for a participant who discontinued from the study.
Measure: Number; unit: Participants
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No
Number analyzed (Participants) | 359 | 368
Participants
  Month 1, >=2 points, n=358, 367 | 225 | 149
  Month 1, >=3 points, n=358, 367 | 182 | 90
  Month 1, >=25 percent, n=358, 367 | 161 | 76
  Month 3, >=2 points, n=359, 368 | 277 | 221
  Month 3, >=3 points, n=359, 368 | 233 | 172
  Month 3, >=25 percent, n= 359, 368 | 218 | 150
  Month 6, >=2 points, n=359, 368 | 277 | 250
  Month 6, >=3 points, n=359, 368 | 245 | 208
  Month 6, >=25 percent, n=359, 368 | 229 | 189
  Month 9, >=2 points, n=359, 368 | 286 | 276
  Month 9, >=3 points, n=359, 368 | 257 | 222
  Month 9, >=25 percent, n=359, 368 | 247 | 207
  Month 12, >=2 points, n=359, 368 | 291 | 273
  Month 12, >=3 points, n=359, 368 | 261 | 229
  Month 12, >=25 percent, n= 359, 368 | 249 | 214
  Month 15, >=2 points, n=359, 368 | 289 | 275
  Month 15, >=3 points, n=359, 368 | 259 | 243
  Month 15, >=25 percent, n=359, 368 | 245 | 231
  Month 18, >=2 points, n=359, 368 | 288 | 268
  Month 18, >=3 points, n=359, 368 | 262 | 229
  Month 18, >=25 percent, 359, 368 | 245 | 212
  Month 21, >=2 points, n=359, 368 | 292 | 274
  Month 21, >=3 points, n=359, 368 | 267 | 237
  Month 21, >=25 percent, n= 359, 368 | 253 | 224
  Month 24, >=2 points, n=359, 368 | 295 | 279
  Month 24, >=3points, n=359, 368 | 277 | 234
  Month 24, >=25 percent, n= 359, 368 | 261 | 221

3. Secondary Outcome: Change From Baseline in the BPH Impact Index (BII) Score at Months 1, 3, 6, 9, 12, 15, 18, 21, and 24 Using the LOCF Approach
Description: The BII is a 4-item questionnaire covering physical discomfort, worry, bother, and impact on usual activities, with a minimum score of 0 (best) and a maximum score (worst) of 13 points. Individual missing questionnaire responses were imputed, as applicable. Change from Baseline in the BII score was summarized by treatment group using the LOCF approach at each scheduled post-Baseline assessment. LOCF analysis involves bringing forward the last non-missing post-Baseline assessment for a participant with missing data and/or for a participant who discontinued from the study. Estimates are based on the adjusted means from the general linear model: Change from Baseline =Treatment + Cluster + Baseline Value. Baseline is defined as the Visit 2 value if it exists; otherwise, it is the latest of all Screening values. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Months 1, 3, 6, 9, 12, 15, 18, 21, and 24
Population: ITT Population. Participants with data available at the specified time point or using LOCF (post-Baseline) were summarized.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No
Number analyzed (Participants) | 359 | 368
Scores on a scale
  Month 1, n=357, 366 | -1.3 (0.11) | -0.4 (0.11)
  Month 3, n=359, 368 | -1.8 (0.11) | -1.0 (0.11)
  Month 6, n=359, 368 | -1.9 (0.11) | -1.3 (0.11)
  Month 9, n=359, 368 | -2.1 (0.11) | -1.5 (0.11)
  Month 12, n=359, 368 | -2.1 (0.12) | -1.5 (0.12)
  Month 15, n=359, 368 | -2.2 (0.12) | -1.5 (0.12)
  Month 18, n=359, 368 | -2.2 (0.12) | -1.4 (0.12)
  Month 21, n=359, 368 | -2.4 (0.12) | -1.6 (0.12)
  Month 24, n=359, 368 | -2.4 (0.12) | -1.6 (0.12)

4. Secondary Outcome: Change From Baseline in the BPH-related Health Status (BHS) Score at Months 1, 3, 6, 9, 12, 15, 18, 21, and 24 Using the LOCF Approach
Description: Each participant was asked the following question "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?". This response was rated from 0 ("delighted") to 6 ("terrible"). Change from Baseline in the BHS score was summarized by treatment group using the LOCF approach at each scheduled post-Baseline assessment. LOCF analysis involves bringing forward the last non-missing post-Baseline assessment for a participant with missing data and/or for a participant who discontinued from the study. Estimates are based on the adjusted means from the general linear model: Change from Baseline =Treatment + Cluster + Baseline Value. Baseline is defined as the Visit 2 value if it exists; otherwise, it is the latest of all Screening values. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Months 1, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No
Number analyzed (Participants) | 359 | 368
Scores on a scale
  Month 1, n=358, 367 | -0.8 (0.06) | -0.3 (0.05)
  Month 3, n=359, 368 | -1.1 (0.06) | -0.7 (0.06)
  Month 6, n=359, 368 | -1.2 (0.06) | -0.9 (0.06)
  Month 9, n=359, 368 | -1.3 (0.06) | -1.0 (0.06)
  Month 12, n=359, 368 | -1.3 (0.06) | -1.1 (0.06)
  Month 15, n=359, 368 | -1.4 (0.06) | -1.1 (0.06)
  Month 18, n=359, 368 | -1.4 (0.06) | -1.1 (0.06)
  Month 21, n=359, 368 | -1.5 (0.06) | -1.1 (0.06)
  Month 24, n=359, 368 | -1.5 (0.06) | -1.1 (0.06)

5. Secondary Outcome: Number of Events of Clinical Progression (CP) of BPH
Description: The number of participants with the first occurrence of clinical progression (CP) of BPH occurring on or after the randomization date are summarized by treatment and year. Time is based on the date of the first-occurring CP event, and is relative to the randomization date. CP of BPH is a composite of five endpoints assessed through the end of the study, including: symptom deterioration by IPSS >=3 points from Baseline (Visit 2); acute urinary retention related to BPH; incontinence (overflow or urge) related to BPH; recurrent urinary tract infection (UTI) or urosepsis related to BPH; renal insufficiency related to BPH (a single >=50% rise from Baseline serum creatinine and a total value >=1.5 milligrams/deciliter). For components that required multiple episodes, the first of the multiple episodes was utilized in terms of timing.
Time Frame: Up to 2 years
Population: ITT Population. Only those participants at risk for CP at the specified visit were analyzed.
Measure: Number; unit: Events
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No
Number analyzed (Participants) | 369 | 373
Events
  Year 1, n=369, 373 | 48 | 94
  Year 2, n=276, 251 | 17 | 14

6. Secondary Outcome: Number of Participants With the Indicated First-occurring Component of Clinical Progression (CP) of BPH
Description: CP of BPH is a composite of five endpoints assessed through the end of the study, including: symptom progression (symptom deterioration by IPSS >=3 points from Baseline [Visit 2]); acute urinary retention (AUR) related to BPH; incontinence (overflow or urge) related to BPH; recurrent urinary tract infection (UTI) or urosepsis related to BPH; renal insufficiency related to BPH (a single >=50% rise from Baseline serum creatinine and a total value >=1.5 milligrams/deciliter). The number of participants with CP of BPH, the number of participants with the indicated first-occurring component of CP of BPH, the number of participants with two simultaneously first-occurring components ("Tied for first component"), and the number of participants with multiple first-occurring components were summarized by treatment group.
Time Frame: Up to Month 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No
Number analyzed (Participants) | 369 | 373
Participants
  Participants with CP of BPH, n=369, 373 | 65 | 108
  BPH symptom progression, n=65, 108 | 59 | 97
  BPH-related AUR, n=65, 108 | 2 | 4
  BPH-related incontinence, n=65, 108 | 4 | 3
  Recurrent BPH-related UTI, n=65, 108 | 0 | 4
  BPH-related renal insufficiency, n=65, 108 | 0 | 0
  Tied for first component, n=65, 108 | 0 | 0
  Multiple components (2 components), n=65, 108 | 4 | 9
  Multiple components (3 components), n=65, 108 | 0 | 1
  Multiple components (>=4 components), n=65, 108 | 0 | 1

7. Secondary Outcome: Number of Participants Who Had Any BPH-related Surgery, Who Had the Indicated Type of Surgery, Who Had 2 BPH-related Surgeries, and Who Had >=3 BPH-related Surgeries
Description: BPH-related surgery was summarized for events occurring on or after the date of randomization. The number of participants who had any BPH-related surgery, the indicated type of surgery, and multiple surgeries was summarized by treatment. Type of surgery data (cystoscopy, transurethral resection of the prostate [TURP], and prostatectomy) are presented in terms of the first-occurring BPH-related surgery after randomization. It was possible for a single participant to have multiple surgeries.
Time Frame: Up to Month 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No
Number analyzed (Participants) | 369 | 373
Participants
  Participants with any BPH-related surgery | 6 | 3
  Participants with cystoscopy | 5 | 1
  Participants with TURP | 2 | 1
  Participants with prostatectomy | 0 | 1
  Participants with 2 surgeries | 1 | 0
  Participants with >=3 surgeries | 0 | 0

8. Secondary Outcome: Number of Participants With the Indicated Responses to Question 1 of the Patient Perception of Study Treatment (PPST) Questionnaire at Baseline and Months 1, 3, 6, 9, 12, 15, 18, 21, and 24 Using the LOCF Approach
Description: The PPST questionnaire consists of two questions (asked to determine how satisfied participants are with the treatment received) and was administered at Baseline and all post-Baseline visits. Question 1 was: "Overall, how satisfied are you with the treatment and its effect on your urinary problems?" There were seven possible responses, including: "very satisfied," "satisfied," "somewhat satisfied," neutral," "somewhat dissatisfied," "dissatisfied," and "very dissatisfied." Response categories were created by grouping together "very satisfied," "satisfied," and "somewhat satisfied" responses into the category of "Any Satisfaction (AS)," and separately grouping "neutral," "somewhat dissatisfied," "dissatisfied," and "very dissatisfied" responses into the category of "Neutral or Any Dissatisfaction (N/AD)." The LOCF method involves bringing forward the last non-missing post-Baseline assessment for a participant with missing data and/or for a participant who discontinued from the study.
Time Frame: Baseline and Months 1, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No
Number analyzed (Participants) | 359 | 364
Participants
  Baseline, Any Satisfaction, n=315, 328 | 119 | 122
  Baseline, Neutral/Any Dissatisfaction, n=315, 328 | 196 | 206
  Month 1, Any Satisfaction, n=358, 349 | 272 | 209
  Month 1, Neutral/Any Dissatisfaction, n=358, 349 | 86 | 140
  Month 3, Any Satisfaction, n= 359, 359 | 300 | 265
  Month 3, Neutral/Any Dissatisfaction, n=359, 359 | 59 | 94
  Month 6, Any Satisfaction, n=359, 361 | 301 | 285
  Month 6, Neutral /Any Dissatisfaction, n=359, 361 | 58 | 76
  Month 9, Any Satisfaction, n=359, 361 | 304 | 293
  Month 9, Neutral/Any Dissatisfaction, n= 359, 361 | 55 | 68
  Month 12, Any Satisfaction, n=359, 363 | 311 | 305
  Month 12, Neutral/Any Dissatisfaction, n=359, 363 | 48 | 58
  Month 15, Any Satisfaction, n=359, 364 | 311 | 299
  Month 15, Neutral/Any Dissatisfaction, n=359, 364 | 48 | 65
  Month 18, Any Satisfaction, n=359, 364 | 305 | 298
  Month 18, Neutral/Any Dissatisfaction, n=359, 364 | 54 | 66
  Month 21, Any Satisfaction, n=359, 364 | 310 | 300
  Month 21, Neutral/Any Dissatisfaction, n=359, 364 | 49 | 64
  Month 24, Any Satisfaction, n=359, 364 | 312 | 312
  Month 24, Neutral/Any Dissatisfaction, n=359, 364 | 47 | 52

9. Secondary Outcome: Number of Participants With the Indicated Responses to Question 2 of the Patient Perception of Study Treatment (PPST) Questionnaire at Baseline and Months 1, 3, 6, 9, 12, 15, 18, 21, and 24 Using the LOCF Approach
Description: The PPST questionnaire consists of two questions (asked to determine how satisfied participants are with the treatment received) and was administered at Baseline and all post-Baseline visits. Question 2 was: "Would you ask your doctor for the treatment you received in this study?" There were three possible responses, including: "Yes," "No," and "Not sure." Response categories included "Yes" and "No or Not Sure," created by grouping together "No" and "Not sure." The LOCF method involves bringing forward the last non-missing post-Baseline assessment for a participant with missing data and/or for a participant who discontinued from the study.
Time Frame: Baseline and Months 1, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No
Number analyzed (Participants) | 359 | 364
Participants
  Baseline, Yes, n=315, 328 | 109 | 103
  Baseline, No or Not Sure, n=315, 328 | 206 | 225
  Month 1, Yes, n=358, 347 | 224 | 166
  Month 1, No or Not Sure, n=358, 347 | 134 | 181
  Month 3, Yes, n=359, 357 | 232 | 207
  Month 3, No or Not Sure, n=359, 357 | 127 | 150
  Month 6, Yes, n=359, 360 | 232 | 227
  Month 6, No or Not Sure, n=359, 360 | 127 | 133
  Month 9, Yes, n=359, 361 | 238 | 231
  Month 9, No or Not Sure, n=359, 361 | 121 | 130
  Month 12, Yes, n=359, 363 | 240 | 229
  Month 12, No or Not Sure, n=359, 363 | 119 | 134
  Month 15, Yes, n=359, 364 | 246 | 239
  Month 15, No or Not Sure, n=359, 364 | 113 | 125
  Month 18, Yes, n=359, 364 | 235 | 236
  Month 18, No or Not Sure, n=359, 364 | 124 | 128
  Month 21, Yes, n=359, 364 | 249 | 234
  Month 21, No or Not Sure, n=359, 364 | 110 | 130
  Month 24, Yes, n=359, 364 | 243 | 236
  Month 24, No or Not Sure, n=359, 364 | 116 | 128

10. Secondary Outcome: Exposure to Study Drug
Description: Study drug exposure (days) = treatment stop date - treatment start date + 1. Participants in the Watchful Waiting Escalated=Yes subgroup could have been escalated to study drug at any time during the study. Therefore, it is possible that participants were exposed to tamsulosin for a shorter length of time than participants in the dutasteride plus tamsulosin group.
Time Frame: Up to 2 years
Population: Treated Subjects Population: all participants starting protocol pharmacological treatment, either dutasteride plus tamsulosin or (escalated to) tamsulosin, as indicated by a nonmissing electronic Case Report Form treatment start date
Measure: Mean (Standard Deviation); unit: days
Groups:
- Watchful Waiting Escalated=Yes: All participants were given lifestyle advice. If any IPSS was the same or greater than the Baseline value at any study visit (post-randomization), participants received tamsulosin 0.4 mg once daily (Watchful Waiting Escalated=Yes). Tamsulosin was continued until the end of the study unless the participant elected to withdraw from the study.
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting Escalated=Yes
Number analyzed (Participants) | 368 | 229
days | 639.8 (215.49) | 566.3 (195.13)

11. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE) Starting Post-randomization
Description: A post-randomization adverse event is defined as an event with an onset on or after the randomization date or with a missing onset date. An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment was exercised in deciding whether reporting was appropriate in other situations. Refer to the general non-serious AE/SAE module for a list of non-serious AEs (occurring at a frequency threshold of >=5%) and SAEs.
Time Frame: Up to 2 years
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No | Watchful Waiting Escalated=Yes
Number analyzed (Participants) | 369 | 373 | 229
Participants
  Any AE | 190 | 119 | 95
  Any SAE | 38 | 25 | 19

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) starting post-randomization (including events with an onset on or after the randomization date or with a missing onset date) were collected (up to 2 years).
Description: SAEs and non-serious AEs are reported for members of the ITT Population.
Groups:
- Watchful Waiting All: Escalated Yes and No: All participants were given lifestyle advice. If any International Prostate Symptom Score (IPSS) was the same or greater than the Baseline value at any study visit (post-randomization), participants received tamsulosin 0.4 mg once daily (Watchful Waiting Escalated=Yes). Tamsulosin was continued until the end of the study unless the participant elected to withdraw from the study.
Arm/Group | Dutasteride Plus Tamsulosin | Watchful Waiting All: Escalated Yes and No | Watchful Waiting Escalated=Yes
Serious Adverse Events (participants affected / at risk) | 38/369 | 25/373 | 19/229
Other Adverse Events (participants affected / at risk) | 43/369 | 13/373 | 12/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dutasteride Plus Tamsulosin (N=369) | Watchful Waiting All: Escalated Yes and No (N=373) | Watchful Waiting Escalated=Yes (N=229)
Atrial fibrillation (Cardiac disorders) | 4 | 2 | 2
Cardiac failure (Cardiac disorders) | 1 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 1
Heart valve incompetence (Cardiac disorders) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2 | 2
Cellulitis (Infections and infestations) | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 2 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Infective exacerbation of chronic obstructive airways (Infections and infestations) | 1 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 1 | 1
Abdominal sepsis (Infections and infestations) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 2 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1 | 1
Transaminases increased (Investigations) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dutasteride Plus Tamsulosin (N=369) | Watchful Waiting All: Escalated Yes and No (N=373) | Watchful Waiting Escalated=Yes (N=229)
Erectile dysfunction (Reproductive system and breast disorders) | 31 | 4 | 3
Retrograde ejaculation (Reproductive system and breast disorders) | 19 | 10 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.